CLINICAL TRIAL: NCT05747209
Title: Prospective Study of an EXErcise Regimen Designed to Improve Functional Mobility, Body Composition, and Strength After Treatment for Breast Cancer
Brief Title: EXErcise Regimen Designed to Improve Functional Mobility, Body Composition, and Strength After Treatment for Breast CA
Acronym: EXERT-BC
Status: Completed | Type: Observational
Sponsor: Colin Champ, MD (Other)
Responsible Party: Sponsor-Investigator, Colin Champ, MD, Director of the AHN CI Exercise Oncology and Resiliency Center, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Organization: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Other Study IDs: EXERT-BC
Record Dates: First submitted 2022-11-02; First posted 2023-02-28 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard High-load resistance training: Standard exercise regimen utilizes a mixture of compound and isolated movements, focusing on compound exercises. The regimen is a typical standard of care resistance training program and sports performance and strength and conditioning facilities. The observed classes will take place three times per week. Warm-up exercises focused on mobility, flexibility and core activation will be performed to reduce the risk of injury. Each individual exercise workout will generally progress from most intense, CKC, compound, and athletic movements to least intense throughout the workout to maximize safety. Additionally, each workout will provide full body resistance training to focus on functional exercises, intensity, and efficiency. Each workout will take approximately 45 minutes. The total exercise regimen will last 3 months.
  Interventions: Other: Observation of Exercise Program Adherence

INTERVENTIONS:
Other: Observation of Exercise Program Adherence — Observation of a monitored group exercise regimen utilizing standard of care high-load resistance training and functional exercises with compound movements under close supervision and with the goal of improving functional mobility, body composition, and strength after cancer treatment to study adherence and attendance to the exercise program.

SUMMARY:
The goal of this clinical trial is to learn how a group resistance training plan can improve body mobility and strength in female breast cancer patients who have completed their breast cancer treatment. The main questions it aims to answer are:

* Is resistance training feasible following breast cancer treatment
* Can it improve the body's mobility and strength lost as a result of the breast cancer treatment
* can it improve the body's composition (for example muscle mass)
* can resistance training increase one's activity level and help prevent weight gain, perhaps, lowering the risk of cancer recurrence.

Participants will attend a group resistance training exercise group program, 3-4 times per week, under close supervision with monitoring a participant's ability to safely and effectively complete the program. The exercises include: lunges, squats and dead lifts.

DETAILED DESCRIPTION:
Obesity and low muscle mass, i.e. poor body composition, is a risk factor for breast cancers and disease recurrence after treatment. Furthermore, weight gain during and after treatment for breast cancer is associated with higher risk of recurrence, distant metastases, and death. Activity levels have been repeatedly associated with a lower risk of cancer incidence, improved outcomes after cancer treatment and improved overall survival, yet the majority of breast cancer survivors do not meet adequate daily activity level recommendations.

This protocol seeks to prospectively follow forty (40) female breast cancer patients (ages 20-95) during exercise who are post-cancer treatment and to assess the safety and feasibility of a monitored group exercise regimen utilizing high-load resistance training and functional exercises with compound movements under close supervision and with the goal of improving functional mobility, body composition, and strength after cancer treatment. This regimen is a standard of care regimen utilized in strength and conditioning protocols. The investigators hypothesize that an observed exercise regimen such as this will prove safe and feasible in women and may improve functional mobility, body composition and resting metabolic rate.

The exercise regimen will utilize a mixture of compound movements utilizing mainly closed kinetic chain movements (CKC), focusing on exercises with the goal of improving physical and metabolic function, mobility, muscle mass and body composition utilizing guidelines from the National Strength and Conditioning Association (NSCA). CKC exercises include lunges, squats, and dead lifts.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-89 years
2. Women with a biopsy proven diagnosis of ductal carcinoma in situ or invasive carcinoma of the breast
3. Women must have undergone breast conservation therapy with no neoadjuvant or adjuvant chemotherapy (adjuvant endocrine therapy is permitted)
4. Participants must have abstained from smoking for at least 12 months
5. Women of child-bearing potential must have had a pregnancy test prior to initiation of radiation therapy (standard protocol for radiation therapy); verbally confirm lack of pregnancy prior to enrollment; and, consent to use adequate contraception during the course of the study.
6. Participants must be determined capable of engaging in resistance training.
7. Participants must have a schedule amenable to three prescheduled workout sessions per week, scheduled during the day.
8. Participants must complete a Functional Mobility Screen (FMS) and be determined safe to engage in the workout regimen by the study exercise personnel.
9. Participants must be determined capable of engaging in group resistance training sessions by exercise personnel and/or study PI
10. Participants must be able to get down and up from the ground and squat their body weight.

Exclusion Criteria:

1. Any treatment with chemotherapy for breast cancer
2. Inability to get and down off the ground or squat body weight
3. Inability to safely engage in group sessions
4. Severe arthritic, joint, cardiovascular, or musculoskeletal condition

Ages: 20 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Females aged 20-89 years with newly diagnosed ductal carcinoma in situ (DCIS) or invasive carcinoma of the breast who have undergone and completed treatment for breast cancer, including one or more of the following: surgery, radiation therapy, chemotherapy, immunotherapy, or hormonal therapy.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Champ, MD, Principal Investigator — AGH Radiation Oncology
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carpenter DJ, Peluso C, Hilton C, Velasquez F, Annichine A, Matsko K, Rosenberg J, Diaz AK, Hyde P, Beriwal S, Champ CE. EXERT-BC: A pilot study of an exercise regimen designed to improve functional mobility, body composition, and strength after the treatment for breast cancer. Cancer Med. 2024 Mar;13(5):e7001. doi: 10.1002/cam4.7001. PMID 38491821

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 54 total patients screened for eligibility (Fig. 2).
  There were 9 patients who chose not to participate due to scheduling conflicts
  There were 2 patients screened who were referred to PT due to joint & musculoskeletal conditions precluding safe training
Period: Overall Study
Arm/Group | Standard High-load Resistance Training
Started | 43
Enrolled Patients Completed the Exercise Regimen and Were Thus Included in Analysis. | 40
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Standard High-load Resistance Training
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 56.5 [51 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Session Attendance
Description: Calculated as the percentage of participants completing at least 75% of the planned exercise sessions. Dropout rate, defined as individuals who quit the workout regimen altogether, is expected to be less 20%.
Time Frame: Baseline and Three (3) months
Population: Participants who completed at least 75% of the planned exercise sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard High-load Resistance Training
Number analyzed (Participants) | 40
Participants | 39

2. Primary Outcome: Change in Adipose Tissue (InBody, kg)
Description: Change in adipose tissue (kg) pre and post resistance training regimen measured via InBody 970 bioelectrical impedance analysis. Values reported are median changes with interquartile range (IQR).
Time Frame: Baseline and Three (3) months
Population: Participants whose change in adipose tissue was measured.
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Standard High-load Resistance Training
Number analyzed (Participants) | 40
kg
  Baseline | 30.7 [21.4 to 40.0]
  Post-Intervention | 28.2 [19.4 to 40.9]

3. Primary Outcome: Change in Adipose Tissue (Ultrasound, Lbs)
Description: Change in adipose tissue (pounds) pre and post resistance training regimen measured via ultrasound. Values reported are median changes with interquartile range (IQR).
Time Frame: Baseline and Three (3) months
Measure: Median (Inter-Quartile Range); unit: percentage of Body Fat
Arm/Group | Standard High-load Resistance Training
Number analyzed (Participants) | 40
percentage of Body Fat
  Baseline | 37.4 [33.0 to 39.6]
  Post-Intervention | 32.6 [28.2 to 37.8]

4. Primary Outcome: Change in Muscle Mass
Description: Changes in percent muscle mass (measured by InBody bioelectrical impedance analysis) from baseline to three months.
Time Frame: Baseline and Three (3) months
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Standard High-load Resistance Training
Number analyzed (Participants) | 40
kg
  InBody Muscle Mass Baseline | 25.0 [23.4 to 27.9]
  InBody Muscle Mass Post-intervention | 25.6 [23.6 to 28.0]

5. Primary Outcome: Change in Fat-Free Mass
Description: Changes in percent fat-free mass (measured by ultrasound) from baseline to three months.
Time Frame: Baseline and Three (3) months
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Standard High-load Resistance Training
Number analyzed (Participants) | 40
kg
  InBody fat Free Mass Baseline | 45.9 [43.0 to 50.4]
  InBody fat Free Mass Post-intervention | 46.9 [43.3 to 50.8]

6. Primary Outcome: Quality of Life Via the EuroQol Group Survey EuroQol-5 Dimensions-5 Levels
Description: EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) test pre and post regimen. This test is a descriptive system that is a preference-based health-related quality of life measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. There is an additional question measuring an individual's current overall health-related quality of life. Total score for the 5 questions ranges from 5 (no problems on any dimension) to 25 (extreme problems on all dimensions). Calculated by assigning scores of 1 (minimum), 2, 3, 4, and 5 (maximum), to the response categories of "no problems", "slight problems", "moderate problems", "severe problems", and "extreme problems"/"unable to", respectively. Higher scores mean worse outcomes. There is an additional question scored from 0 to 100 recorded for their current overall health-related quality of life. 100 means the best health and 0 means the worst health they can imagine.
Time Frame: Baseline and Three (3) months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard High-load Resistance Training
Number analyzed (Participants) | 40
score on a scale
  EuroQol 5 Dimension 1: Mobility Score Baseline | 5 [5 to 5]
  EuroQol 5 Dimension 1: Mobility Score Post-Intervention | 5 [5 to 5]
  EuroQol 5 Dimension 2 Self-Care Score Baseline | 5 [5 to 5]
  EuroQol 5 Dimension 2 Self-Care Score Post-Intervention | 5 [5 to 5]
  EuroQol 5 Dimension 3 Usual Activities Score Baseline | 5 [5 to 5]
  EuroQol 5 Dimension 3 Usual Activities Score Post-Intervention | 5 [5 to 5]
  EuroQol 5 Dimension 4 Pain / Discomfort Score Baseline | 4 [4 to 5]
  EuroQol 5 Dimension 4 Pain / Discomfort Score Post-Intervention | 4 [4 to 5]
  EuroQol 5 Dimension 5 Anxiety / Depression Score Baseline | 5 [4 to 5]
  EuroQol 5 Dimension 5 Anxiety / Depression Score Post-Intervention | 5 [4.8 to 5]
  EuroQol 5 Dimension 6 Current Overall Health-Related Quality of Life Score Baseline | 73.5 [60 to 86.3]
  EuroQol 5 Dimension 6 Current Overall Health-Related Quality of Life Score Post-Intervention | 85 [70 to 95]

7. Primary Outcome: Activity Levels Via Godin Questionnaire
Description: Change in activity levels measured by Godin Questionnaire pre and post regimen, specifically strenuous, moderate and mild/light exercise with a score from 0 to unlimited. The Godin scale score lists 24 or more units of exercise as active, 14-23 units as moderately active, and less than 14 units as insufficiently active/sedentary
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard High-load Resistance Training
Number analyzed (Participants) | 40
score on a scale
  Baseline | 23.5 [6 to 35.3]
  Post-intervention | 41.5 [32.8 to 55.5]

8. Primary Outcome: Resting Metabolic Rate as Calories Burned Per Day
Description: Change in resting metabolic rate (RMR) pre and post regimen measured via ultrasound and bioimpedance analysis.
Time Frame: Baseline and Three (3) months
Measure: Median (Inter-Quartile Range); unit: kcal
Arm/Group | Standard High-load Resistance Training
Number analyzed (Participants) | 40
kcal
  InBody RMR Baseline | 1365.5 [1305.5 to 1453.8]
  InBody RMR Post-intervention | 1381.5 [1306.3 to 1467.3]
  US RMR Baseline | 1403 [1324 to 1482.8]
  US RMR Post-intervention | 1437 [1352.3 to 1540]

9. Primary Outcome: Functional Movement Screen
Description: A functional movement screen will be performed pre and post regimen to assess change in overall score
  Functional movement screen (FMS) total score for the 7 movement patterns assessed by an examiner ranges from 0 to 21. A score below 14 is felt to identify individuals at risk of injury. This is calculated by assigning scores of 0 (minimum), 1, 2, and 3 (maximum) to the response categories of "if any pain felt by the subject during the movement", "subject is unable to perform the movement", "subject performs the movement through compensatory movements", and "subject performs the movement correctly", respectively. A score below 14 is felt to identify individuals at risk of injury. Higher scores mean a better outcome.
Time Frame: Baseline and Three (3) months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard High-load Resistance Training
Number analyzed (Participants) | 40
score on a scale
  Baseline | 9 [8 to 11]
  Post-intervention | 12 [9.8 to 14]

10. Primary Outcome: Y-balance Score
Description: A Y-balance test will be performed pre and post regimen to assess change
  Y-balance score adds up the distance each leg can move in the front and side directions, divided by the length of the hip. This correlates inversely with fall risk.
Time Frame: Baseline and Three (3) months
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Standard High-load Resistance Training
Number analyzed (Participants) | 40
ratio
  Baseline Left Side | 72.3 [63.9 to 81.2]
  Post-intervention Left Side | 83.9 [78.3 to 98.1]
  Baseline Right Side | 73.0 [62.3 to 80.2]
  Post-intervention Right Side | 86.2 [76.5 to 95.0]

11. Primary Outcome: Changes in Strength From Baseline Through Study Completion, up to 3 Months
Description: Strength will be calculated via load lifted throughout the entire regimen as weight x repetitions x sets at the end of months 1, 2, and 3.
Time Frame: Baseline and months 1, 2, and 3
Measure: Median (Inter-Quartile Range); unit: Load (kilograms x Repetitions x Sets)
Arm/Group | Standard High-load Resistance Training
Number analyzed (Participants) | 40
Load (kilograms x Repetitions x Sets)
  Load Split Squat, Month 1 (Week 4) | 192 [15 to 299]
  Load Split Squat, Month 2 (Week 4) | 383 [268 to 479]
  Load Split Squat, Month 3 (Week 4) | 383 [327 to 585]
  Load Trap Bar Deadlift, Month 1 (Week 4) | 1131 [912 to 1298]
  Load Trap Bar Deadlift, Month 2 (Week 4) | 1210 [944 to 1527]
  Load Trap Bar Deadlift, Month 3 (Week 4) | 1415 [1012 to 1667]
  Incline Dumbbell Bench, Month 1 (Week 4) | 170 [136 to 204]
  Incline Dumbbell Bench, Month 2 (Week 4) | 261 [204 to 278]
  Incline Dumbbell Bench, Month 3 (Week 4) | 272 [265 to 352]
  Bird Dog Row, Month 1 (Week 4) | 204 [136 to 228]
  Bird Dog Row, Month 2 (Week 4) | 272 [204 to 310]
  Bird Dog Row, Month 3 (Week 4) | 340 [299 to 374]

12. Secondary Outcome: Participants Will Undergo an Assessment 1 Year Following the Exercise Program.
Description: Participants will be assessed 1 year following exercises as they were at baseline and post exercise as Standard of Care (SOC). The SOC assessments will encompass weight, height, BMI, body composition, resting metabolic rate, quality of life questionnaires and exercise forms, strength, and mobility
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months per patient
Description: AEs/SAEs meet the ct.gov definitions: accidental disclosure of confidentiality and injury from exercise program All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were monitored/assessed, but none were observed.
Arm/Group | Standard High-load Resistance Training
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT05747209/Prot_SAP_000.pdf